CLINICAL TRIAL: NCT01381926
Title: Changes in Bone Turnover With Exposure to a GLP-1 Receptor Agonist (UAB Core Center for Basic Skeletal Research)
Brief Title: Changes in Bone Turnover With Exposure to a GLP-1 Receptor Agonist
Acronym: CMBD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unavailability of study drug and matching placebo
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Principal Investigator, Amy H. Warriner, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F100929001
Record Dates: First submitted 2011-06-13; First posted 2011-06-27 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus; Bone Remodeling
Keywords: Type 2 diabetes; exenatide; Byetta
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Exenatide then Placebo (Experimental): Study participants in phase1 will receive the study drug, exenatide, at a dose of 5mg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of exenatide will be increased to 10mg subcutaneously twice daily before meals for one month. During the third month of the study, no study medication will be given and this will serve as a "wash out" period prior to the second phase of the study (placebo). During the fourth and fifth months, study participants will get placebo alternatives to exenatide 5mg and exenatide 10mg, respectively, subcutaneously twice daily before meals.
  Interventions: Drug: exenatide; Drug: Saline
- Placebo then Exenatide (Active Comparator): Study participants in phase1 will receive the saline placebo, at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the saline placebo will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no treatment will be given and this will serve as a "wash out" period prior to the second phase of the study. During the fourth month study participants will receive Exenatide 5mcg twice daily with meals. During the fifth month, study participants will receive exenatide 10mcg, subcutaneously twice daily before meals.
  Interventions: Drug: exenatide; Drug: Saline

INTERVENTIONS:
Drug: exenatide — exenatide 5mcg sq twice daily for one month and exenatide 10mcg twice daily for month 2. The 3rd month is a washout period. Month 4 and 5 saline placebo is given as 5mcg and 10mcg respectively.
  Other Names: Byetta
Drug: Saline — Month 1 and 2 saline placebo is given as a low and high dose respectively. The 3rd month is a washout period. Month 4 exenatide 5mcg sq twice daily and for month 5 exenatide 10mcg twice daily is administered.
  Other Names: Normal Saline

SUMMARY:
The purpose of this study is to determine changes in bone turnover markers and calcitonin following the initiation of exenatide compared to placebo in postmenopausal women wtih type 2 diabetes.

Hypothesis 1a: Bone resorption (measured by osteocalcin and bone-specific alkaline phosphatase) will be lower and bone formation (measured by type I collagen crosslinked aminoterminal peptide in urine (Urine NTX)) will be higher when subjects are treated with exenatide compared to when subjects are treated with placebo.

Hypothesis 1b: Calcitonin levels will not vary significantly between periods of treatment with exenatide vs. placebo.

DETAILED DESCRIPTION:
Patients with Type 2 Diabetes Mellitus (T2DM) are at an increased risk of fracture, despite having bone mineral density (BMD) levels similar to age and sex matched cohorts. Recent studies have indicated that changes in incretin (INtestinal seCRETion of INsulin) hormones in the setting of T2DM may play a role in bone metabolism. Two of these incretin hormones, gastric inhibitory polypeptide (GIP) and glucagon-like peptide-1 (GLP-1), have been shown to be involved in bone turnover regulation, in addition to their effect in increasing insulin secretion and decreasing glucagon secretion in a glucose-dependent manner. In addition, the rise in glucagon-like peptide-2 (GLP-2) in the postprandial state has been found to have a direct effect on reduced bone resorption in a non-fasting state and treatment with GLP-2 improved BMD in postmenopausal women. Due to their glucose lowering effects, incretin hormones have been a therapeutic target for the treatment of T2DM through GLP-1 receptor agonists (i.e. exenatide) or inhibition of incretin hormone metabolism via dipeptidyl peptidase 4 (DPP-4)inhibitors. The GLP-1 receptor analog exenatide leads to an approximate 13-fold increased GLP-1 effect compared to approximate doubling of incretin hormone levels with current DDP-4 inhibitors. In rodent models, calcitonin levels rise significantly following treatment with GLP-1 receptor agonists, leading to c-cell hyperplasia. However, review of calcitonin changes in humans and cynomolgus monkeys treated with GLP-1 receptor agonists have not shown similar results.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (as defined by age ≥45 years old or amenorrhea for >2years)
* Type 2 DM currently not on diabetes-specific medication(s) or treated with monotherapy of metformin or a sulfonylurea. Patients treated with insulin monotherapy will also be eligible if the total daily dose of insulin is ≤10units. If on a medication for diabetes prior to study entry, the medication can be discontinued for 2 weeks prior to study initiation.
* Hemoglobin A1c (HbA1c) of 6.5-9.0%

Exclusion Criteria:

* Use of an incretin mimetic (i.e. exenatide, liraglutide), a DPP-4 inhibitor (i.e. sitagliptin, saxagliptin), a thiazolidinedione, or oral glucocorticoids in the 6 months prior to the study will not be eligible
* Known osteoporosis or patients treated with an osteoporosis-specific medication (bisphosphonate, teriparatide) or estrogen (including Selective Estrogen Receptor Modulators (SERMs)) or those who anticipate imminent treatment with one of these medications will be excluded from the study
* Chronic kidney disease (calculated GFR <30 ml/min) or a disease known to affect bone turnover (i.e. Paget Disease, Osteogenesis Imperfecta, HIV) will be excluded from the study.
* History of pancreatitis

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Warriner, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol open to accrual: February 2011, primary completion date, August 2015 and study completion date August 2015. Recruitment location at UAB. Postmenopausal women with diabetes mellitus on no medications or metformin alone were recruited from a single outpatient clinic setting.
Pre-assignment Details: Potential participants attended a screening visit to ensure they met inclusion/exclusion criteria. If they were on metformin at the screening visit, it was discontinued. They returned in 1 month for the baseline visit and randomization.
Groups:
- Exenatide 1st Then Placebo: Study participants in period 1 will receive the study drug, exenatide, at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of exenatide will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no study medication will be given and this will serve as a "wash out" period prior to the second period of the study (placebo). During the fourth and fifth months, study participants will get placebo alternatives to exenatide 5mcg and exenatide 10mcg, respectively, subcutaneously twice daily before meals.
- Placebo 1st Then Exenatide: Study participants in periods1 will receive the saline placebo at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of saline placebo will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no treatment will be given and this will serve as a "wash out" period prior to the second periods of the study. During the fourth month participants will receive Exenatide 5mcg twice daily before meals. During the fifth month, study participants will get Exenatide 10mcg twice daily before meals.
Period: Low/High Dose of 1st Treatment (2months)
Arm/Group | Exenatide 1st Then Placebo | Placebo 1st Then Exenatide
Started (The number of participants started is for each segment. Crossover study. Total is not applicable.) | 5 | 5
Completed | 3 | 4
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Low/High Dose of 2nd Treatment (2months)
Arm/Group | Exenatide 1st Then Placebo | Placebo 1st Then Exenatide
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study. Not all patients completed both arms of the study. 14 patients were screened. 10 presented for the baseline study and were provided some study medication. 1 participant's specimen was not analyzed and she is not included in analysis for that reason. 5 started Exenatide; 5 started Placebo.
Groups:
- Placebo 1st Then Exenatide: Study participants in period1 will receive the saline placebo at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of saline placebo will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no treatment will be given and this will serve as a "wash out" period prior to the second periods of the study. During the fourth month participants will receive Exenatide 5mcg twice daily before meals. During the fifth month, study participants will get Exenatide 10mcg twice daily before meals.
- Total: Total of all reporting groups
Arm/Group | Placebo 1st Then Exenatide | Exenatide 1st Then Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (4.2) | 61 (3.8) | 61 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Determine Changes in Bone Resorption Markers During the Treatment With a GLP-1 Receptor Agonist (Exenatide) Compared to Placebo in Patients With T2DM.
Description: Bone reabsorption by bone-specific alkaline phosphatase (BAP) was assessed. Distribution of the Difference between EX/PBO Low/High Dose and Baseline Levels were calculated.
Time Frame: Baseline to 20 weeks
Population: For Crossover study, participants were matched for the placebo and study drug arms. As such, only data from participants completing both arms were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Exenatide 1st Then Placebo: Study participants in phase1 will receive the study drug, exenatide, at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of exenatide will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no study medication will be given and this will serve as a "wash out" period prior to the second phase of the study (placebo). During the fourth and fifth months, study participants will get placebo alternatives to exenatide 5mcg and exenatide 10mcg, respectively, subcutaneously twice daily before meals.
- Placebo 1st Then Exenatide: Study participants in phase1 will receive the saline placebo at a dose of 5mcg subcutaneously twice daily 30 minutes before meals for one month. During the second month of the study, the dose of saline placebo will be increased to 10mcg subcutaneously twice daily before meals for one month. During the third month of the study, no treatment will be given and this will serve as a "wash out" period prior to the second phase of the study. During the fourth month participants will receive Exenatide 5mcg twice daily before meals. During the fifth month, study participants will get Exenatide 10mcg twice daily before meals.
Arm/Group | Exenatide 1st Then Placebo | Placebo 1st Then Exenatide
Number analyzed (Participants) | 3 | 4
mg/L | 1.925 (1.6) | -0.20 (3.34)

2. Primary Outcome: Determine Changes in Bone Turnover Markers by Serum N-Telo Peptide During the Treatment With a GLP-1 Receptor Agonist (Exenatide) Compared to Placebo in Patients With T2DM.
Description: Bone turnover by Serum N-Telo peptide (NTX) was assessed. Distribution of the Difference between EX/PBO Low/High Dose and Baseline Levels were calculated
Time Frame: Baseline to 20 weeks
Population: For Crossover, study, participants were matched for the placebo and study drug arms. As such, only data from participants completing both arms were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: nMBCE/L
Arm/Group | Exenatide Then Placebo | Placebo Then Exenatide
Number analyzed (Participants) | 3 | 4
nMBCE/L | -0.8 (2.31) | 1.725 (2.72)

3. Primary Outcome: Determine Changes in Bone Turnover Markers by Tartrate-Resistant Acid Phosphatase 5b (TRACP5b) During the Treatment With a GLP-1 Receptor Agonist (Exenatide) Compared to Placebo in Patients With T2DM.
Description: Bone turnover by Tartrate-Resistant Acid Phosphatase 5b (TRACP5b) was assessed. Distribution of the Difference between EX/PBO Low/High Dose and Baseline Levels were calculated.
Time Frame: Baseline to 20 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Exenatide 1st Then Placebo | Placebo 1st Then Exenatide
Number analyzed (Participants) | 3 | 4
U/L | 0.05 (0.80) | 0.325 (0.59)

ADVERSE EVENTS:
Time Frame: Baseline to 20 weeks
Description: clinicaltrials.gov definitions used
Arm/Group | Exenatide 1st Then Placebo | Placebo 1st Then Exenatide
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide 1st Then Placebo (N=3) | Placebo 1st Then Exenatide (N=4)
Nausea/vomiting (1st treatment period) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritis (2nd treatment period) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was closed due to unavailability of study drug/matching placebo prior to recruitment of target participants. The original drug company was bought and new company was unwilling to supply medication. Small participant number limits data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No